CLINICAL TRIAL: NCT04690504
Title: Proteomic and Transcriptomic Biomarkers of Circadian Timing - Validation of Circadian Biomarkers in Patients With Sleep Disorders
Brief Title: Validation of Circadian Biomarkers in Patients With Sleep Disorders
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Jeanne Duffy, Co-Investigator, Brigham and Women's Hospital
Other Study IDs: 2020-P-000606
Record Dates: First submitted 2020-12-15; First posted 2020-12-30 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Sleep Disorders, Circadian Rhythm; Circadian Rhythm Disorders; Circadian Rhythm Sleep Disorder; Advanced Sleep Phase Syndrome (ASPS); Delayed Sleep Phase Syndrome; Sleep Wake Disorders; Sleep Disorder
Keywords: ASWPD, DSWPD, CRSWD, melatonin, circadian, circadian rhythm, biomarker
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Chronobiology Disorders; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples will be collected and assayed for melatonin. Blood samples will be collected and assayed for rhythmic gene transcripts and rhythmic proteins. A blood sample will be collected for DNA analysis, including potential GWAS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dim light melatonin onset (DLMO) — A series of saliva samples will be collected and assayed for melatonin so that the timing of melatonin secretion onset can be determined.

SUMMARY:
Current methods for assessing circadian timing require sampling over hours (or even up to a day) while the patient is in controlled conditions. The investigators aim to develop a method that can estimate individual circadian time with a single blood sample taken at any time of the day or night. To do this, the investigators will use two state of the art methods, a plasma proteomics-based method to identify a panel of rhythmic proteins (extending our preliminary data) and a whole blood-derived monocyte-based method using a panel of 15 transcripts (to validate and extend a recent study).

We will test both methods in a series of patients with circadian rhythm sleep disorders. We will validate separately the proteomics-based biomarker and the monocyte-based transcript biomarker, and also explore whether combining them can improve the accuracy of our timing estimates. In all cases, circadian phase estimates from the biomarker panels will be compared with those derived from plasma or saliva melatonin (the current "gold-standard" circadian phase marker).

DETAILED DESCRIPTION:
Adults who meet ICSD-3 criteria for Advanced Sleep Wake Phase Disorder or Delayed Sleep Wake Phase Disorder will be studied at Brigham and Women's Hospital and Stanford University.

The outpatient protocol will consist of two segments: clinic visit and in-home saliva sample collection. For the first segment, the patient participant will be scheduled for a daytime visit to the sleep clinic where they will have blood drawn for protein and monocyte analysis after having kept a sleep diary and worn a wrist activity monitor for at least 1 week. The patient participant will be provided with an at-home saliva sampling kit and instructed in its use, in particular how to maintain appropriate dim light conditions. For the second segment, the patient will be instructed to collect the series of saliva samples on that same evening, collecting a saliva sample each hour beginning 7 hours before their usual bedtime and ending one hour after their usual bedtime. As each sample is collected, the patient participant will document the tube number and clock time on a log that the investigators provide them, and the patient participant will store each sample in a zip lock bag in their home freezer until the next day. After waking the next day, the patient will pack their samples in the insulated shipping box they were provided, along with their sample collection log and freezer packs they were provided, and then they call a courier to pick up the box, which is sent directly to the assay facility.

Alternatively, patients may be given the opportunity to come for a single extended visit at the laboratory or clinic. This visit will include the blood sampling for protein and monocyte analysis, followed by 8 hours in which they remain in dim lighting conditions in the lab or clinic and provide a saliva sample each hour. The saliva sampling segment will begin 7 hours before their usual bedtime and ending one hour after their usual bedtime. After the final saliva sample the study will be over and the patient will be allowed to go home.

ELIGIBILITY:
Inclusion Criteria:

* ICSD3 diagnosis of Advanced Sleep-Wake Phase Disorder or Delayed Sleep-Wake Phase Disorder
* otherwise healthy

Exclusion Criteria:

* history of drug or alcohol dependency
* a sleep disorder other than a circadian rhythm sleep disorder
* use of medications that interfere with melatonin production (e.g., beta blockers) within the past month
* night shift work (for ASWPD patients) or early morning starts (for DSWPD patients) in the prior 3 years
* recent (within 3 months) travel to a place 2 time zones or greater away from home
* acute or uncontrolled medical conditions
* major visual deficit
* active or uncontrolled psychological or psychiatric disorder
* use of exogenous melatonin or melatonin agonists within the past month

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy adults who meet ICSD-3 criteria for Advanced Sleep Wake Phase Disorder (ASWPD) or Delayed Sleep Wake Phase Disorder (DSWPD).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
DLMO | Study Day 1
  dim light melatonin onset, the time at which melatonin levels in the saliva rise above 3pg/mL
BodyTime | Study Day 1
  the time at which a series of rhythmic gene transcripts predict circadian phase
PlasmaTime | Study Day 1
  the time at which a series of rhythmic proteins predict circadian phase

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Mignot, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No